CLINICAL TRIAL: NCT06610890
Title: Pharmacokinetic Interactions Between Hemay005 Tablets and Midazolam Maleate Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM005PS1S08
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Hemay005; Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy subject (Experimental): Midazolam maleate tablets 15 mg were taken orally in the morning on Day1, and Hemay005 tablets were taken daily on Day3-Day9, twice a day, 60mg once. Midazolam maleate tablets 15 mg+Hemay005 tablets 60mg were taken orally in the morning of Day10
  Interventions: Drug: Hemay005; Drug: Midazolam maleate

INTERVENTIONS:
Drug: Hemay005 — One 15mg tablet, four tablets at a time
  Other Names: Hemay005 tablet
Drug: Midazolam maleate — One 15mg tablet, one tablet at a time
  Other Names: Midazolam maleate tablet

SUMMARY:
1. To evaluate the pharmacokinetics of Hemay005 tablets on midazolam and its active metabolite α-hydroxymidazolam after multiple administration;
2. Evaluate the effect of Hemay005 tablet on QT interval;
3. To investigate the effect of Hemay 005 tablets on inflammatory factors.

DETAILED DESCRIPTION:
1. To evaluate the pharmacokinetics of Hemay005 tablets on midazolam and its active metabolite α-hydroxymidazolam after multiple administration;
2. Evaluate the effect of Hemay005 tablet on QT interval;
3. To investigate the effect of Hemay 005 tablets on inflammatory factors.
4. The safety of the subjects was evaluated

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged from 18 to 65 years old (including 18 and 65 years old), the ratio of male to female was 1:1;
* Body weight: male ≥50.0kg, female ≥45.0kg, body mass index [BMI= weight (kg)/height 2 (m2)] between 19.0 kg/m2 and 26.0kg/m2 (including boundary values);
* 90mmHg≤ systolic blood pressure <140mmHg, 60mmHg≤ diastolic blood pressure <90 mmHg, 60 beats/min ≤ pulse ≤100 beats/min, normal body temperature (abnormal vital signs could be retested, normal retest results were considered to meet the inclusion criteria);
* The results of ECG were normal or abnormal but not clinically significant, including QTcF≤450 ms in men and QTcF≤470 ms in women, PR interval

  * 200ms and QRS complex duration ≤110 ms;
* Before the trial, they have understood the nature, significance, possible benefits, possible inconvenience and potential risks of the trial in detail, and voluntarily participate in the clinical trial, can communicate well with the investigators, comply with the requirements of the whole study, and sign the written informed consent.

Exclusion Criteria:

* those who participated in other drug clinical trials within 3 months;
* patients with abnormal clinical manifestations that need to be excluded, including but not limited to diseases of the nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal system, respiratory system, metabolic system, skeletal system and other systems, especially patients with myasthenia gravis, schizophrenia and severe depression;
* patients with any disease that increases the risk of bleeding, such as active or previous history of gastrointestinal ulcer, gastrointestinal bleeding or perforation, ulcerative colitis, or intracranial hemorrhage;
* a history of vomiting, diarrhea, or any physiological condition that could interfere with the test results within 7 days before the test;
* those with a history of specific allergies (asthma, urticaria, eczema, etc.), or allergic to any drug, food or pollen, or known allergic to Hemay 005, midazolam or other benzodiazepines;
* those who have lost or donated more than 400mL of blood within 3 months before the trial, or intend to donate blood during the trial;
* Pregnant or lactating women, or subjects (including male subjects) have plans to have children or to donate sperm or eggs from two weeks before the study to three months after the last dose of the study, and are unwilling or unable to take effective contraceptive measures;
* general physical examination and laboratory tests (blood routine, blood biochemistry, coagulation function, urine routine, stool routine, blood β-human chorionic gonadotropin/urine pregnancy (female), etc.) within 7 days before the test, chest X-ray within 1 month before the test, and electrocardiogram (ECG) within 14 days before the test judged by clinicians to be clinically significant;
* persons with one or more positive results of hepatitis B surface antigen, hepatitis C virus antibody, HIV antigen antibody or syphilis specific antibody;
* patients with clinically significant major diseases or major surgical procedures within 3 months before the trial;
* drank more than 14 units of alcohol per week (1 unit = 17.7 mL ethanol, i.e. 1 unit = 357 mL of 5% beer or 43 mL of 40% liquor or 147 mL of 12% wine) in the 3 months before the trial, or could not abstain from alcohol during the trial;
* who smoked more than 5 cigarettes per day in the 3 months before the trial, or who could not stop using any tobacco products during the trial;
* consuming excessive amounts of tea, coffee and/or caffeine-rich beverages (> 8 cups, 1 cup =250 mL) per day in the 3 months before the trial;
* consuming any foods or drinks (such as strong tea, coffee, chocolate, cola, animal organs, grapefruit, dragon fruit, mango, etc.) rich in caffeine/xanthine or other special ingredients (such as strong tea, coffee, chocolate, cola, animal organs, grapefruit, dragon fruit, mango, etc.) from screening to -2 days of admission, or unable to stop eating the above foods or drinks during the trial;
* use of any drugs (e.g., inducers - barbiturates, carbamazepine, phenytoin, glucocorticoids) that inhibit or induce hepatic drug-metabolizing enzymes within 30 days before the test; Inhibitors (SSRI antidepressants, cimetidine, sedative-hypnotics, verapamil, fluoroquinolones, antihistamines);
* those who are unable to eat or have dysphagia, have special dietary requirements and/or cannot follow a uniform diet;
* patients with a history of asthma or seizures;
* who used any prescription medication, over-the-counter medication, nutrine, herbal medicine product or received a vaccination within 14 days before the trial; Or plan to take non-trial drugs or supplements during the trial; Or use of a drug for less than 5 half-lives before taking the study drug, whichever is longer;
* Mechanical operators engaged in high-altitude work, motor vehicle driving and other dangerous operations;
* those who cannot tolerate venipuncture and/or have a history of dizzy with blood or needles;
* had used any drug in the past year;
* alcohol breath test results > 0.0mg/100mL or drug abuse screening positive (morphine, methamphetamines, ketamine, dimethylenedioxyamphetamine, tetrahydrocannabinol acid, cocaine);
* Subjects who were considered by the investigator to have poor adherence or any factor that precluded participation in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Relevant pharmacokinetic parameters，Peak Plasma Concentration（Cmax） | Day1-Day12
  All subjects who receive the drug will be analyzed for pharmacokinetic
Relevant pharmacokinetic parameters，Area under the plasma concentration versus time curve（AUC0-t） | Day1-Day12
  All subjects who receive the drug will be analyzed for pharmacokinetic
Relevant pharmacokinetic parameters，Area under the curve from time 0 extrapolated to infinite time (AUC0-inf) | Day1-Day12
  All subjects who receive the drug will be analyzed for pharmacokinetic

SECONDARY OUTCOMES:
QT interval | Day1，Day3-9
  All subjects who receive the drug will be analyzed for QT interval
Detection of inflammatory factors | Day1，Day9
  The concentrations of certain cytokines were determined，for example： CRP (C-reactive protein), Haptoglobin (haptoglobin), Fibrinogen (fibrinogen), albumin (albumin), IL-6 (interleukin-6), TNF-α (tumor necrosis factor-α), MCP-1 (monocyte chemoattractant protein-1), MCP-3 (McP-3). Monocyte chemoattractant protein-3 (McT-3), calprotectin, CD11b and CD66b .

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China